CLINICAL TRIAL: NCT06530849
Title: A Phase 1/2 Clinical Study of GC012F Injection in Subjects With Refractory Systemic Lupus Erythematosus
Brief Title: A Study of GC012F Injection in Subjects With Refractory Systemic Lupus Erythematosus
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Gracell Biotechnologies (Shanghai) Co., Ltd. (Industry)
Collaborators: AstraZeneca (Industry); Suzhou Gracell Biotechnologies Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D8313C00002
Record Dates: First submitted 2024-07-25; First posted 2024-07-31 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Refractory Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GC012F Injection (Experimental): GC012F Injection
  Interventions: Drug: GC012F Injection

INTERVENTIONS:
Drug: GC012F Injection — GC012F Injection is an autologous chimeric antigen receptor T cell therapy targeting both BCMA and CD19

SUMMARY:
This is a single-arm, open-label, multicenter, phase 1/2 clinical study to assess the safety and efficacy of GC012F Injection in subjects with refractory Systemic Lupus Erythematosus (SLE).

DETAILED DESCRIPTION:
This is a single-arm, open-label, multicenter, phase 1/2 clinical study to assess the safety and efficacy of GC012F Injection in subjects with refractory SLE；The dose-escalation phase 1 study aims to assess the safety of GC012F Injection and determine the Recommended Phase II Dose (RP2D). The phase 2 study aims to determine the efficacy and safety of GC012F Injection at the RP2D in patients with refractory SLE and assess the pharmacokinetics (PK) and pharmacodynamics (PD) characteristics.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the ICF;
2. Males or females, aged 18-70 years old (inclusive);
3. Must be able and willing to comply with the study visit schedule and other protocol requirements;
4. Presence of CD19+B cells in the peripheral blood;
5. Diagnosed with SLE and meeting the 2019 EULAR/ACR classification criteria for SLE;
6. Used standard SLE treatment regimens and at least a biological agent for more than 6 months but did not meet the LLDAS criteria
7. SLEDAI-2000 scores ≥8 during the screening period. If the scores for low complement and/or anti-ds-DNA antibody are available, the SLEDAI-2000 scores for clinical symptoms (except low complement and/or anti-ds-DNA antibody) should be NLT 4;
8. Positive serological test results of autoantibodies: Positive results of antinuclear antibody (ANA) and/or anti-ds-DNA antibody and/or anti-Sm antibody, with critical values not acceptable;
9. Adequate functional reserve of organs:

   1. Neutrophil count ≥1 × 10^9/L, lymphocyte count ≥0.3 × 10^9/L; hemoglobin ≥85 g/L; platelet count ≥50 × 10^9/L;
   2. ALT ≤3 × ULN; AST ≤3 × ULN; TBIL ≤2 × ULN;
   3. Creatinine clearance ≥40 mL/min;
   4. Left ventricular ejection fraction (LVEF) ≥45% and no pericardial effusion with clinical significance as diagnosed by echocardiography; no abnormal ECG with clinical significance;
   5. Oxygen saturation ≥92%; no pleural effusion with clinical significance.
10. Females of childbearing potential must:

    1. Have a negative serum β-hCG pregnancy test confirmed by investigators during the screening period;
    2. Agree and be able to use effective contraceptives continuously from the screening to at least 1 year after the infusion of GC012F Injection. Contraceptive methods must include one highly effective method and one additional effective (barrier) method, which should be used from the screening until at least 1 year after the infusion of GC012F Injection or until absence of CAR-T cells shown by two consecutive qPCR assays (whichever occurs later);
    3. Agree to avoid breastfeeding during the study period until at least 1 year after the infusion of GC012F Injection or until absence of CAR-T cells shown by two consecutive quantitative polymerase chain reaction (qPCR) assays (whichever occurs later);
11. Male subjects must agree to use condoms during sexual contact with pregnant females or females of childbearing potential for at least 1 year after the infusion of GC012F Injection, even if a successful vasectomy has been performed;
12. Venous access available for blood collection, and no contraindications for leukapheresis.

Exclusion Criteria:

1. Receipt of CD19 and/or BCMA-targeted therapies or CAR T-cell therapies for any targets in the past;
2. Receipt of CD20-targeted drug therapy within 6 months prior to screening;
3. Receipt of immunosuppressants or prednisone >15 mg/d or equivalent doses of other glucocorticoids within 1 week before the apheresis;
4. Presence of any renal disorders: serious lupus nephritis (serum creatinine >2.5 mg/dL or 221 μmol/L), or active nephritis requiring treatments with drugs forbidden in this protocol, or any needs for hemodialysis within 8 weeks prior to apheresis;
5. Presence of any serious heart diseases as follows:

   1. Congestive heart failure (New York Heart Association (NYHA) Class III or IV);
   2. Myocardial infarction or receipt of coronary artery bypass grafting (CABG) within 6 months prior to screening;
   3. Clinically significant ventricular arrhythmias or a history of unexplained syncope not due to vasovagal reaction or dehydration; or a QTc interval >480 ms during the screening;
   4. A medical history of severe non-ischemic cardiomyopathy;
6. Need for supplemental oxygen or mechanical ventilation with oxygen saturation <92%;
7. Hypertension uncontrolled by drug therapies;
8. A medical history of any central nervous system (CNS) or neurodegenerative diseases due to or not due to SLE
9. Clinically significant hemorrhage symptoms or definite bleeding tendencies (such as gastrointestinal bleeding and bleeding gastric ulcer), hereditary or acquired bleeding and thrombophilia (such as hemophilia, coagulation disorder, and hypersplenism) within 3 months prior to screening; arteriovenous thrombosis events, such as cerebrovascular diseases (including cerebral hemorrhage and cerebral infarction), deep vein thrombosis, and/or pulmonary embolism within 6 months prior to screening;
10. Any history of active malignancy or malignancy within 5 years prior to screening. The following circumstances should be excluded: early-stage tumors that have received radical treatment (carcinoma in situ or grade 1 tumors, or non-ulcerative primary melanoma with a depth <1 mm and no involvement of lymph nodes), basal cell carcinoma, squamous cell carcinoma, cervical carcinoma in situ, or breast cancer in situ that has received potential radical treatment;
11. Immunodeficiency, active viral or bacterial infection (requiring systemic antimicrobial therapy) or uncontrolled systemic fungal infection;
12. Any positive results of the following items: Human immunodeficiency virus (HIV) antibody positive; HBsAg positive; or HBcAb positive (subjects with HBV DNA copy numbers below the lower limit of detection can be enrolled); hepatitis C antibody (HCV-Ab) positive (the subjects with HCV RNA below the lower limit of detection can be enrolled) or a known medical history of hepatitis C; treponema pallidum antibody (TP-Ab) positive;
13. Receipt of a live-attenuated vaccine within 4 weeks prior to apheresis;
14. A history of severe hypersensitivity or allergy;
15. Contraindication or hypersensitivity to fludarabine, cyclophosphamide, and any component of the investigational product;
16. Receipt of surgeries within 2 weeks prior to apheresis or a plan to receive surgeries during the study (except for a plan of local anesthesia surgery, which should not be performed within 2 weeks after infusion);
17. Pregnant women or lactating women who do not agree to abstain from breastfeeding, and men and women who have a fertility plan during the participation in this study or within 1 year after receiving the study treatment;
18. Participation in any other clinical trials within 4 weeks prior to signing the informed consent form, or the date of signing the informed consent form still within 5 half-lives of the last dose of the drug of the last clinical trial (whichever is longer);
19. Any situations that may hinder the participation of the subjects in the entire trial or confound the results, or any situations in which investigators believe that the participation in this study is not in the best interests of the subjects.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-08-22 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity (DLT) rate | 28 days
  Phase 1 study：Proportions of subjects with DLT within 28 days after infusion.
SLE Responder Index (SRI)-4 response rate | 48 weeks
  Phase 2 study：Proportion of subjects achieving SRI-4 response at Week 48.

SECONDARY OUTCOMES:
adverse events (AEs) | 48 weeks
  Proportions of subjects with AEs after the infusion;
SRI-4 response rate | 48 weeks
  Proportions of subjects achieving SLE Responder Index (SRI)-4 response by timepoint;
Definitions of Remission in SLE (DORIS) rate | 48 weeks
  Proportions of subjects achieving remission according to the DORIS by timepoint;
lupus low disease activity state (LLDAS) rate | 48 weeks
  Proportions of subjects achieving LLDAS by timepoint;
complete remission (CR) rate | 48 weeks
  Proportions of subjects achieving CR by timepoint;
SRI-4 response duration | 48 weeks
  Maintenance time of SRI-4 response;
DORIS duration | 48 weeks
  Maintenance time of remission according to the DORIS;
LLDAS duration | 48 weeks
  Maintenance time of LLDAS;
CR duration | 48 weeks
  Maintenance time of complete remission

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Research Site, Shanghai
  - Research Site, Wuhan